CLINICAL TRIAL: NCT05578755
Title: Evaluation of a Novel Intervention Aimed at Instilling Future-oriented Mindsets and Behaviors Using a Smartphone Application and Immersive Virtual Reality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Responsible Party: Principal Investigator, Jean-Louis van Gelder, Professor, Universiteit Leiden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 772911-CRIMETIME
Record Dates: First submitted 2022-10-05; First posted 2022-10-13 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Future Orientation; Self-defeating Behavior; Future Self-identification
Keywords: Smartphone application; Virtual reality; Digital behavior change intervention; Future self-identification; Future orientation; Self-defeating behavior; Goals; Short-term mindsets; Long-term mindsets; Intervention; Randomized Controlled Trial; Engagement
MeSH Terms: interventions — Organizational Objectives

STUDY DESIGN:
Intervention Model Description: There are three arms: 1) smartphone-based intervention, 2) immersive virtual reality intervention, and 3) active, goal-setting, control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smartphone-based intervention (Experimental)
  Interventions: Behavioral: FutureU
- Virtual reality intervention (Experimental)
  Interventions: Behavioral: FutureU
- Goal-setting control condition (Active Comparator)
  Interventions: Behavioral: Goal-setting

INTERVENTIONS:
Behavioral: FutureU — FutureU is based on the assumption that future orientation can be strengthened by increasing the extent to which people identify with their future self. People who identify more with their future self appear to be more inclined to make more altruistic choices favoring their future self and foregoing immediate gratification. The intervention provides psychoeducation and exposure to and interaction with the future self. Participants interact with a digitally aged version of themselves, i.e., their 'future self', using a smartphone application (app) or through immersive virtual reality (VR).
  The app consists of three week-long modules. Participants interact with the app on a daily basis for about 5 minutes a day for 21 consecutive days.
  The VR consists of three sessions, each lasting about 30 minutes. Each VR session is guided by a trained researcher.
  Arms: Smartphone-based intervention; Virtual reality intervention
Behavioral: Goal-setting — In the control condition participants set goals (as in the intervention conditions), but receive no further guidance.
  Arms: Goal-setting control condition

SUMMARY:
Short-term thinking, or the inability to make informed tradeoffs between immediate benefits and longer-term costs, has been related to a variety of negative or self-defeating behaviors, such as substance use, impulsive decision making, and delinquency, whereas future-oriented thinking tends to be positively associated with positive behaviors, such as self-esteem, planning, and goal-directed behaviors. To bolster people's psychosocial development, the investigators are developing an intervention, FutureU, aimed at instilling future-oriented mindsets and behaviors by strengthening people's identification with who they may be in the future, i.e., their 'future self'. Through the use of a smartphone application (app) and immersive virtual reality (VR), participants interact with a visual representation of their future self. In the present study, the investigators will evaluate the current iteration of this intervention and compare the FutureU app and FutureU VR with each other and with a goal-setting control group. Knowledge and insights gained from this study will be used to further develop the FutureU intervention program and can provide insights for intervention theory building and implementation strategies.

DETAILED DESCRIPTION:
People with a short-term mindset tend be focused on the here-and-now and are inclined to disregard the more distant consequences of their actions. This often results in self-defeating behaviors, i.e., behaviors that provide immediate gains but that may simultaneously incur significant costs in the longer run (e.g., substance use, delinquency, overspending). In contrast, people who are more future-oriented typically balance the immediate gains against the longer-term consequences of their decisions and are more inclined to set goals for the future. The investigators are developing an intervention, FutureU, aiming to promote future-oriented mindsets and behaviors by strengthening people's identification with their 'future self'. The level of identification with the future self depends on the extent to which people are able to vividly imagine their future self (i.e., vividness), feel positively towards their future self (i.e., valence), and feel similar and connected to their future self (i.e., related). During the intervention, participants interact with their future self. This future self is developed on the basis of a digitally aged image of themselves. In order to present the visual representation of the participants' future self, the investigators implement the intervention via a smartphone application (app) and via immersive virtual reality (VR). The present study examines the current iteration of the FutureU intervention, which is developed within an ongoing research program. The findings of this study will be used to further develop and optimize the FutureU intervention.

In a three-armed Randomized Controlled Trial, the investigators will evaluate the FutureU intervention by examining 1) its effectiveness on both proximal and distal outcomes, 2) its working mechanisms, and 3) moderators of intervention effects. It is hypothesized that FutureU will increase participants' future-oriented mindsets and behaviors (e.g., increase future orientation, enhance goal achievement, and reduce self-defeating behaviors). There are no specific expectations regarding differences in effectiveness between the two implementation strategies (app vs. VR). Regarding the working mechanisms, the hypothesis is that intervention effects of FutureU are mediated by increases in future self-identification. Concerning moderators, the investigators will examine the moderating role of personality traits within an intervention context in an exploratory fashion. Furthermore, associations between usage patterns (e.g., length and frequency of use), engagement levels and intervention outcomes will be examined, and the goals set by the participants will be analyzed qualitatively and quantitatively.

ELIGIBILITY:
Inclusion Criteria:

* First-year university student
* Dutch speaking

Exclusion Criteria:

* Epileptic symptoms (due to VR condition)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Future self-identification | Change from baseline to 6-months follow-up (assessed at baseline, 1 and 2 weeks after baseline (i.e., during the intervention), 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Future self-identification, that is, the degree to which people have a clear image of their future self and can identify with their future self, will be assessed with 8 items based on Hershfield et al. (2009) and Van Gelder et al. (2015). These items measure the degree to which people can imagine their future self vividly (i.e., vividness), the level of positive feelings towards the future self (i.e., valence), and the extent to which people feel connected and similar to their future self (i.e., relatedness).
Future Orientation | Change from baseline to 6-months follow-up (assessed at baseline, 1 and 2 weeks after baseline (i.e., during the intervention), 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Future orientation measuring time perspective, anticipation of future consequences, and planning ahead will be assessed with the Future orientation Scale (Steinberg et al., 2009) consisting of 15 items (α = .80).
Consideration of future consequences | Change from baseline to 6-months follow-up (assessed at baseline, 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  The degree to which people take immediate versus distant consequences into account in potential behaviors will be assessed with the Consideration of Future Consequences questionnaire (Bruderer Enzler, 2013; Strathman et al., 1994) consisting of 9 items.
Self-defeating behavior | Change from baseline to 6-months follow-up (assessed at baseline, 1 and 2 weeks after baseline (i.e., during the intervention), 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Self-defeating behavior, that is, behaviors with immediate gains though long-term costs, will be measured with 15 items representing different self-defeating behaviors based on the measure of Van Gelder et al. (2015).
Goal commitment | Change from baseline to 6-months follow-up (assessed at baseline, 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Commitment to the goal participants set for the year will be measured using the Goal Commitment Questionnaire (Hollenbeck et al., 1989) which consists of 7 items (α = .71).
Goal achievement | Assessed during the 3-week intervention.
  Weekly and monthly goal achievement will be assessed with 3 self-developed items measuring how often participants thought about their goal, worked towards their goal, and to what extend they achieved their goal.

SECONDARY OUTCOMES:
Self-efficacy | Change from baseline to 6-months follow-up (assessed at baseline, 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Self-efficacy, that is, people's sense of competence to effectively deal with life stressors, will be measured with the General Self-efficacy Questionnaire (Schwarzer & Jerusalem, 1995) consisting of 10 items (range α = .75 - .91).
Academic results | Up to 10 months after baseline
  Academic results, i.e., grade point average, will be requested from the university at the end of the academic year after participants' consent.
Impulsiveness | Change from baseline to 6-months follow-up (assessed at baseline, 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  Impulsiveness, indicated by lack of impulse control on planning, motor, and attention will be assessed with the Barratt Impulsiveness Scale short form (Spinella, 2007) consisting of 15 items (α = .79).

OTHER OUTCOMES:
Thinking about the future | Change from baseline to 6-months follow-up (assessed at baseline, 1 and 2 weeks after baseline (i.e., during the intervention), 3 weeks after baseline (i.e., post measurement), and 3- and 6-months follow-up)
  We will ask participants how often in the past week they thought about their future and their future self (2 items).
Personality | Assessed at baseline and 6-months follow-up.
  Personality will be measured with the Dutch version of the 60-item HEXACO-PI-R (Lee & Asthon, 2018). This questionnaire measures 6 personality dimensions: Honesty-Humility, Emotionality, Extraversion, Agreeableness, Conscientiousness, and Openness to Experience. Dimensions are assessed with 10 items each (range α = .82 - .89).
Users' engagement and log data of the smartphone application | Assessed during the 3-week intervention.
  In the FutureU app condition, we use the nine-item TWente Engagement with Ehealth Technologies Scale (TWEETS) to measure users' engagement with the app (range α = .86 - .87). We measure engagement with the app's specific features (e.g., opinion regarding the avatar appearance, and specific modules) with self-developed items. Participants' usage patterns are captured in the app its log-data (e.g., number of days the app was opened and time spent in the app).
Users' engagement and log data of the FutureU immersive virtual reality | Assessed during the 3-week intervention.
  In the FutureU VR condition, we measure users' experiences within and of the VR (e.g., embodiment, presence, and appearance avatar) and participants' (objective) behavioral data in VR (e.g., total time spent in the VR environment, number of switches between avatars, what questions they ask their future self).
Participants' goals | Assessed during the 3-week intervention.
  Qualitative assessment of the goals participants set at the start and during the intervention, measuring aspects such as goal specificity, goal difficulty, topic of the goal, and goal type.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis van Gelder, Prof.dr.dr., Principal Investigator — Max Planck Institute for the Study of Crime, Security, and Law; Leiden University
Locations (1):
- Leiden University, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mertens ECA, Siezenga AM, Tettero T, van Gelder JL. A future orientation intervention delivered through a smartphone application and virtual reality: study protocol for a randomized controlled trial. BMC Psychol. 2022 Dec 20;10(1):315. doi: 10.1186/s40359-022-01025-x. PMID 36539846